CLINICAL TRIAL: NCT00896389
Title: The Relationship Between Serine Threonine Kinase 39 (STK39) Genotypes, Salt Sensitivity, Thiazide Diuretics-induced Blood Pressure Response
Brief Title: Salt Loading and Thiazide Intervention Study
Acronym: SALTI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Yen-Pei Christy Chang, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040712; R21DK084566 (NIH)
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2018-05-31 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Hypertension
Keywords: hypertension; hydrochlorothiazide; HCTZ; Salt sensitivity; Hydrochlorothiazide induced hyperglycemia
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Salt-loading and thiazide diuretic (HCTZ) (Other): Salt loading:2 L of 0.9% NaCl. HCTZ:12.5/ 25 mg of HCTZ for 1 week
  Interventions: Procedure: Salt loading; Drug: Hydrochlorothiazide (HCTZ)

INTERVENTIONS:
Procedure: Salt loading — Subjects will arrive at the Amish Research Clinics after overnight fasting. After taking height, weight, BP, and body temperature, subjects will receive 2 liters (L) of 0.9% sodium chloride (NaCl) saline over 4 hours while their blood pressure is monitored every 15 minutes. Blood pressure will be taken every 15 minutes during this procedure. Blood and urine samples will be collected from all subjects pre- and post-infusion.
Drug: Hydrochlorothiazide (HCTZ) — We will perform short-term HCTZ intervention on the same 120 subjects. After overnight fasting and having their height, weight, and BP measured, subjects are given seven 12.5 mg HCTZ tablets and instructed to take 1 tablet daily for one week. Ambulatory blood pressure will be measured and blood and urine will be collected on both day 1 and day 8. After a minimum 6-week wash-out period, the subjects will repeat the 7-day HCTZ intervention, taking 25 mg of HCTZ instead. Subjects with plasma potassium levels below 3.6 mmol/L on day 8 of 12.5 mg HCTZ will be given a daily supplement of 16 milliequivalents of potassium to prevent harmful loss of potassium while taking HCTZ.
  Other Names: Hydrochlorothiazide; HCTZ; Apo-Hydro; Aquazide H; Dichlotride; Hydrodiuril; HydroSaluric; Microzide; Esidrex; Oretic.

SUMMARY:
The investigators of this study propose to examine the relationships between STK39 (Serine Threonine Kinase 39) genotypes and responses to salt loading and to thiazide diuretics, hydrochlorothiazide. The investigators hypothesize that STK39 genotypes will be associated with the outcome of both interventions and can contribute to personalized care for hypertension.

DETAILED DESCRIPTION:
Although hypertension can be easily diagnosed and there are many medications available to treat hypertension, this condition is poorly managed in many patients and is a leading cause of morbidity and mortality worldwide. Because a newly identified hypertension susceptibility gene, STK39 (Serine Threonine Kinase 39), plays a central role in kidney sodium transport, the investigators propose a pharmacogenetics study to examine the relationships between STK39 genotypes and blood pressure responses to salt loading and to thiazide diuretics, hydrochlorothiazide. In addition, STK39 genotypes may also predict those hypertension patients more likely to develop thiazide-induced hyperglycemia. The investigators hypothesize that STK39 genotypes of those single nucleotide polymorphisms (SNPs) that are associated with baseline systolic blood pressure (SBP), diastolic blood pressure (DBP), and hypertension status, will be associated with the outcome of both interventions. Therefore these SNPs can act as markers and contribute to personalized care for hypertension by identifying patients most likely to effectively control their blood pressure by adopting salt-reducing diet versus patients most likely to effectively and safely control their blood pressure by taking thiazide diuretics.

ELIGIBILITY:
Inclusion Criteria:

* Old Order Amish
* Age 18 to 65
* Have systolic blood pressure between 120 and 160 and diastolic blood pressure between 80 and 100

Exclusion Criteria:

* History of myocardial infarction, stroke, congestive heart failure, liver disease
* Known cause of secondary hypertension
* Diabetes or Fasting glucose > 100 mg/dL
* Women who are pregnant, on oral contraceptives, or menstruating
* Used hydrochlorothiazide (HCTZ) in the last 8 weeks or known allergy to HCTZ
* Taking non-steroidal anti-inflammatory drugs
* Estimated glomerular filtration rate < 80 mL/m
* Intention to alter dietary habit during the study
* Abuse of alcohol or drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yen Pei C. Chang, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Amish Research Clinics, Lancaster, Pennsylvania, United States

REFERENCES:
- [Background] Wang Y, O'Connell JR, McArdle PF, Wade JB, Dorff SE, Shah SJ, Shi X, Pan L, Rampersaud E, Shen H, Kim JD, Subramanya AR, Steinle NI, Parsa A, Ober CC, Welling PA, Chakravarti A, Weder AB, Cooper RS, Mitchell BD, Shuldiner AR, Chang YP. From the Cover: Whole-genome association study identifies STK39 as a hypertension susceptibility gene. Proc Natl Acad Sci U S A. 2009 Jan 6;106(1):226-31. doi: 10.1073/pnas.0808358106. Epub 2008 Dec 29. PMID 19114657
- [Background] Delpire E, Gagnon KB. SPAK and OSR1: STE20 kinases involved in the regulation of ion homoeostasis and volume control in mammalian cells. Biochem J. 2008 Jan 15;409(2):321-31. doi: 10.1042/BJ20071324. PMID 18092945
- [Background] Chiga M, Rai T, Yang SS, Ohta A, Takizawa T, Sasaki S, Uchida S. Dietary salt regulates the phosphorylation of OSR1/SPAK kinases and the sodium chloride cotransporter through aldosterone. Kidney Int. 2008 Dec;74(11):1403-9. doi: 10.1038/ki.2008.451. Epub 2008 Sep 17. PMID 18800028

RESULTS

PARTICIPANT FLOW:
Groups:
- Salt-loading and Thiazide Diuretics (HCTZ): Salt loading: 2 liters (L) of 0.9% sodium chloride (NaCl). HCTZ:12.5 or 25 mg of HCTZ for 1 week
Period: Salt Loading
Arm/Group | Salt-loading and Thiazide Diuretics (HCTZ)
Started | 124
Completed | 124
Not Completed | 0
Period: HCTZ Low Dose
Arm/Group | Salt-loading and Thiazide Diuretics (HCTZ)
Started | 28 (Only subjects with SBP > 120 mmHg and agreeable to the HCTZ protocol continued to the next period.)
Completed | 28
Not Completed | 0
Period: HCTZ High Dose
Arm/Group | Salt-loading and Thiazide Diuretics (HCTZ)
Started (Of the 28 subjects that started HCTZ intervention, 3 terminated the study without completing.) | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Salt-loading and Thiazide Diuretic (HCTZ): Salt loading: Subjects will arrive at the Amish Research Clinics after overnight fasting. After taking height, weight, BP, and body temperature, subjects will receive 2 L of 0.9% NaCl (sodium chloride) saline over 4 hours while their blood pressure is monitored every 15 minutes. Blood pressure will be taken every 15 minutes during this procedure. Blood and urine samples will be collected from all subjects pre- and post-infusion.
  Hydrochlorothiazide (HCTZ): After overnight fasting and having their height, weight, and BP measured, subjects are given 12.5 mg HCTZ tablets and instructed to take 1 tablet daily for one week. Ambulatory blood pressure, blood and urine will be collected on both day 1 and day 8. After a wash-out period, the subjects will repeat the HCTZ intervention, taking 25 mg HCTZ instead.
Arm/Group | Salt-loading and Thiazide Diuretic (HCTZ)
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Only subjects whose baseline blood pressure is high enough (SBP>120 or DBP>80 mmHg) and willing to undergo the multi-week intervention were enrolled into the HCTZ part of the study.
  years
    Saline infusion only | 50 (7)
    saline infusion and HCTZ: number analyzed (Participants) | 28
    saline infusion and HCTZ | 53 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 53
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Only subjects whose baseline blood pressure is high enough (SBP>120 or DBP>80 mmHg) and willing to undergo the multi-week intervention were enrolled into the HCTZ part of the study.
  mmHg
    Salt loading | 114 (11)
    HCTZ: number analyzed (Participants) | 28
    HCTZ | 126 (10)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Only subjects whose baseline blood pressure is high enough (SBP>120 or DBP>80 mmHg) and willing to undergo the multi-week intervention were enrolled into the HCTZ part of the study.
  mmHg
    Salt Loading | 71 (7)
    HCTZ: number analyzed (Participants) | 28
    HCTZ | 80 (7)
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.1 (2.8)
creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.74 (0.12)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Change During Salt Loading
Description: Systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured every 15 minutes for 4 hours.
  Blood pressure change is calculated by the trapezoid method. Essentially we use the average of blood pressure at each pair of time points (for example, DBP 30min + DBP 15min)/2 + (DBP 45min + DBP 30min)/2 + … up to 4 hours.) normalized by baseline SBP/DBP.
Time Frame: Every 15 minutes for 4 hours
Population: 124 subjects were divided into 3 genotype groups based on their rs35929607 genotypes. Genotype GG is homozygous for the minor allele G, genotype AG is heterozygous, and genotype AA is homozygous for the major allele A.
Measure: Mean (Standard Error); unit: mmHg
Groups:
- rs35929607 SNP: Single nucleotide polymorphism (SNP) rs35929607, located in an intron of serine threonine kinase 39 (STK39) gene, is associated with blood pressure in the Amish population.
  This SNP, rs35929607, has 2 alleles, A and G. Allele G is found less frequently and has an allele frequency of approximately 0.2-0.4 in populations studied thus far. We genotyped all participants of this study and determine if they are homozygous for the G allele, i.e., have the GG genotype, or are heterozygous (AG genotype), or are homozygous for the A allele and have the AA genotype.
Arm/Group | rs35929607 SNP
Number analyzed (Participants) | 124
mmHg
  DBP, Genotype GG: number analyzed (Participants) | 2
  DBP, Genotype GG | -25.5 (4.3)
  DBP, Genotype AG: number analyzed (Participants) | 32
  DBP, Genotype AG | 34.6 (11.6)
  DBP, Genotype AA: number analyzed (Participants) | 90
  DBP, Genotype AA | 23.2 (7.7)
  SBP, Genotype GG: number analyzed (Participants) | 2
  SBP, Genotype GG | -41.4 (8.4)
  SBP, Genotype AG: number analyzed (Participants) | 32
  SBP, Genotype AG | 62.9 (15.7)
  SBP, Genotype AA: number analyzed (Participants) | 90
  SBP, Genotype AA | 44.8 (10.6)
Statistical Analysis 1: Comparison: rs35929607 SNP; Null hypothesis: There is no association between STK39 SNP rs35929607 genotype group and phenotypes collected in this study; Test type: Other — Association between genotypes and phenotypes were tested using a linear mixed model, coding genotype as an independent variable with an additive genetic effect, and including age, age^2, and sex as covariates in the model. All association analyses were run using the Mixed Models for Pedigree Analysis (MMAP) software program to account for the relatedness among study subjects. MMAP User Guide is available from http://edn.som.umaryland.edu/mmap/index.php; p > 0.05, Chi-squared — Because no P-values less than 0.05 was observed, we did not adjust them for multiple comparison to avoid false positives

2. Secondary Outcome: Change in Plasma Aldosterone Level Due to Salt-loading
Description: Aldosterone is a hormone that plays a critical role in homeostatic regulation of blood pressure. Change is defined as the post-salt loading values minus the pre-salt loading values
Time Frame: Aldosterone was measured from blood collected pre and post salt loading
Population: 124 subjects were divided into 3 genotype groups based on their rs35929607 genotypes. Genotype GG is homozygous for the minor allele G, genotype AG is heterozygous, genotype AA is homozygous for the major allele A.
Measure: Mean (Standard Error); unit: ng/dL
Groups:
- rs35929607 SNP: SNP rs35929607, located in an intron of STK39 gene, is associated with blood pressure in the Amish population.
  This SNP, rs35929607, has 2 alleles, A and G. Allele G is found less frequently and has an allele frequency of approximately 0.2-0.4 in populations studied thus far. We genotyped all participants of this study and determine if they are homozygous for the G allele, i.e., have the GG genotype, or are heterozygous (AG genotype), or are homozygous for the A allele and have the AA genotype.
Arm/Group | rs35929607 SNP
Number analyzed (Participants) | 124
ng/dL
  Genotype GG: number analyzed (Participants) | 2
  Genotype GG | -7.5 (4.5)
  Genotype AG: number analyzed (Participants) | 32
  Genotype AG | -1.2 (0.7)
  Genotype AA: number analyzed (Participants) | 90
  Genotype AA | -1.9 (0.6)
Statistical Analysis 1: Comparison: rs35929607 SNP; Test type: Other — Association between genotype and phenotype were tested using a linear mixed model, coding genotype as an independent variable with an additive genetic effect, and including age, age^2, and sex as covariates in the model. All association analyses were run using the Mixed Models for Pedigree Analysis (MMAP) software program to account for the relatedness among study subjects. MMAP User Guide is available from http://edn.som.umaryland.edu/mmap/index.php; p < 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change in Plasma Renin Activity Due to Salt-loading
Description: Renin is an enzyme that mediates extracellular fluid and regulates blood pressure. Plasma renin activity (PRA) is a measure of the activity of the plasma enzyme renin. PRA is measured in the laboratory by incubating plasma at physiologic temperature in a buffer that facilitates its enzymatic activity. The natural substrate for the enzyme renin is angiotensinogen. Exogenous angiotensinogen is not added to the reaction mixture. This means that, in effect, the PRA results reported are dependent on both renin concentration and the concentration of its substrate in the patient's plasma. Renin cleaves angiotensinogen to produce a decapeptide, angiotensin I, the concentration of which is assayed using liquid chromatography accompanied by tandem mass spectroscopic detection (LC/MS/MS). PRA levels are reported as the amount of angiotensin I generated per unit of time. Change is defined as the post-salt loading values minus the pre-salt loading values
Time Frame: Renin was measured from blood collected pre and post salt loading
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/ml/h
Arm/Group | rs35929607 SNP
Number analyzed (Participants) | 124
ng/ml/h
  Genotype GG: number analyzed (Participants) | 2
  Genotype GG | -0.8 (0.3)
  Genotype AG: number analyzed (Participants) | 32
  Genotype AG | -0.3 (0.1)
  Genotype AA: number analyzed (Participants) | 90
  Genotype AA | -0.4 (0.1)
Statistical Analysis 1: Comparison: rs35929607 SNP; Null hypothesis: There is no association between STK39 SNP rs35909607 genotype group and phenotypes collected in this study; Test type: Other — [test comment as in outcome 2, analysis 1]; p > 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change in Plasma Sodium/Potassium Level Due to Salt-loading
Description: Na/K ratio is a function of kidney function
Time Frame: Plasma sodium and potassium measured from blood collected pre and post salt loading
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ratio
Arm/Group | rs35929607 SNP
Number analyzed (Participants) | 124
ratio
  Genotype GG: number analyzed (Participants) | 2
  Genotype GG | 0.3 (0.8)
  Genotype AG: number analyzed (Participants) | 32
  Genotype AG | -0.3 (0.4)
  Genotype AA: number analyzed (Participants) | 90
  Genotype AA | 0.1 (0.2)
Statistical Analysis 1: Comparison: rs35929607 SNP; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p > 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change in Plasma Sodium/Potassium Level During Low Dose of HCTZ
Description: Na/K ratio is a function of kidney function
Time Frame: Plasma sodium and potassium measured from blood collected pre and post salt loading
Population: 28 subjects were divided into 3 genotype groups based on their rs35929607 genotypes. Genotype 11 is homozygous for the minor allele G, genotype 12 is heterozygous, genotype 22 is homozygous for the major allele A.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | rs35929607 SNP
Number analyzed (Participants) | 28
ratio
  Genotype GG: number analyzed (Participants) | 1
  Genotype GG | 0 (0)
  Genotype AG: number analyzed (Participants) | 7
  Genotype AG | 1.0 (0.6)
  Genotype AA: number analyzed (Participants) | 20
  Genotype AA | 0.6 (0.4)
Statistical Analysis 1: Comparison: rs35929607 SNP; [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p > 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

6. Primary Outcome: Blood Pressure Change After 7 Days of Low Dose (12.5 mg) of HCTZ
Description: Blood pressure change is defined as SBP or DBP average over the 24 hour period, Day 8 subtracts Day 0.
Time Frame: 24-hr Ambulatory blood pressure were measured every hour on day 0 and day 8
Population: 28 subjects were divided into 3 genotype groups based on their rs35929607 genotypes. Genotype GG is homozygous for the minor allele G, genotype AG is heterozygous, genotype AA is homozygous for the major allele A.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | rs35929607 SNP
Number analyzed (Participants) | 28
mmHg
  DBP, Genotype GG: number analyzed (Participants) | 1
  DBP, Genotype GG | 0 (0)
  DBP, Genotype AG: number analyzed (Participants) | 7
  DBP, Genotype AG | 2.0 (2.4)
  DBP, Genotype AA: number analyzed (Participants) | 20
  DBP, Genotype AA | -1.1 (1.1)
  SBP, Genotype GG: number analyzed (Participants) | 1
  SBP, Genotype GG | 1.0 (0)
  SBP, Genotype AG: number analyzed (Participants) | 7
  SBP, Genotype AG | -0.7 (4.3)
  SBP, Genotype AA: number analyzed (Participants) | 20
  SBP, Genotype AA | -4.2 (1.3)
Statistical Analysis 1: Comparison: rs35929607 SNP; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p > 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

7. Primary Outcome: Blood Pressure Change After 7 Days of High Dose (25 mg) of HCTZ
Description: Blood pressure change is defined as SBP or DBP average over the 24 hour period, Day 8 subtracts Day 0.
Time Frame: 24-hr Ambulatory blood pressure were measured every hour on day 0 and day 8
Population: 25 subjects were divided into 3 genotype groups based on their rs35929607 genotypes. Genotype GG is homozygous for the minor allele G, genotype AG is heterozygous, genotype AA is homozygous for the major allele A.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | rs35929607 SNP
Number analyzed (Participants) | 25
mmHg
  DBP, Genotype GG: number analyzed (Participants) | 1
  DBP, Genotype GG | -2 (0)
  DBP, Genotype AG: number analyzed (Participants) | 6
  DBP, Genotype AG | 0.7 (2.4)
  DBP, Genotype AA: number analyzed (Participants) | 18
  DBP, Genotype AA | -1.7 (1.1)
  SBP, Genotype GG: number analyzed (Participants) | 1
  SBP, Genotype GG | 1 (0)
  SBP, Genotype AG: number analyzed (Participants) | 6
  SBP, Genotype AG | -1.3 (4.2)
  SBP, Genotype AA: number analyzed (Participants) | 18
  SBP, Genotype AA | -4.5 (1.3)
Statistical Analysis 1: Comparison: rs35929607 SNP; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p > 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

8. Primary Outcome: Fasting Glucose Change After 7 Days of Low Dose (12.5 mg) of HCTZ
Description: Values on Day 8 subtracts Day 0.
Time Frame: Fasting glucose was measured on day 0 and day 8
Population: as for outcome 6
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | rs35929607 SNP
Number analyzed (Participants) | 28
mmHg
  Fasting glucose, GG Genotype: number analyzed (Participants) | 1
  Fasting glucose, GG Genotype | 9 (0)
  Fasting glucose, AG Genotype: number analyzed (Participants) | 7
  Fasting glucose, AG Genotype | 2 (2.5)
  Fasting glucose, AA Genotype: number analyzed (Participants) | 20
  Fasting glucose, AA Genotype | -0.1 (1.2)
Statistical Analysis 1: Comparison: rs35929607 SNP; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p > 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

9. Primary Outcome: Fasting Glucose Change After 7 Days of High Dose (25mg) of HCTZ
Description: Values on Day 8 subtracts Day 0.
Time Frame: Fasting glucose was measured on day 0 and day 8
Population: 25 subjects were divided into 3 genotype groups based on their rs35929607 genotypes. Genotype 11 is homozygous for the minor allele G, genotype 12 is heterozygous, genotype 22 is homozygous for the major allele A.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | rs35929607 SNP
Number analyzed (Participants) | 25
mmHg
  Fasting glucose, GG Genotype: number analyzed (Participants) | 1
  Fasting glucose, GG Genotype | 1.0 (0)
  Fasting glucose, AG Genotype: number analyzed (Participants) | 6
  Fasting glucose, AG Genotype | 1.0 (2.3)
  Fasting glucose, AA Genotype: number analyzed (Participants) | 18
  Fasting glucose, AA Genotype | 2.3 (2.1)
Statistical Analysis 1: Comparison: rs35929607 SNP; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p > 0.05, Chi-squared — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change in Plasma Sodium/Potassium Level During High Dose of HCTZ
Description: Na/K ratio is a function of kidney function
Time Frame: Plasma sodium and potassium measured from blood collected pre and post salt loading
Population: as for outcome 7
Measure: Mean (Standard Error); unit: ratio
Arm/Group | rs35929607 SNP
Number analyzed (Participants) | 25
ratio
  Genotype GG: number analyzed (Participants) | 1
  Genotype GG | 1 (0)
  Genotype AG: number analyzed (Participants) | 6
  Genotype AG | 0 (2.3)
  Genotype AA: number analyzed (Participants) | 18
  Genotype AA | 2.3 (2.1)
Statistical Analysis 1: Comparison: rs35929607 SNP; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p > 0.05, Chi-squared; Because no P-values less than 0.05 was observed, we did not adjust them for multiple comparison to avoid false positives

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Groups:
- Salt Loading: Subjects will arrive at the Amish Research Clinics after overnight fasting. After taking height, weight, BP, and body temperature, subjects will receive 2 L of 0.9% NaCl (sodium chloride) saline over 4 hours while their blood pressure is monitored every 15 minutes. Blood pressure will be taken every 15 minutes during this procedure. Blood and urine samples will be collected from all subjects pre- and post-infusion.
- HCTZ: After overnight fasting and having their height, weight, and BP measured, subjects are given seven 12.5 mg HCTZ tablets and instructed to take 1 tablet daily for one week. Ambulatory blood pressure will be measured and blood and urine will be collected on both day 1 and day 8. After a minimum 6-week wash-out period, the subjects will repeat the 7-day HCTZ intervention, taking 25 mg of HCTZ instead. Subjects with plasma potassium levels below 3.6 mmol/L on day 8 of 12.5 mg HCTZ will be given a daily supplement of 16 milliequivalents of potassium to prevent harmful loss of potassium while taking HCTZ.
Arm/Group | Salt Loading | HCTZ
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/28
Other Adverse Events (participants affected / at risk) | 0/124 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No